CLINICAL TRIAL: NCT02869477
Title: Institut Paoli Calmettes Cardia Cancer Database
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: BDD-CARDIA-IPC
Record Dates: First submitted 2016-08-11; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Stomach Neoplasms; Cardia
MeSH Terms: conditions — Stomach Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with cardia cancer diagnosis
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection

SUMMARY:
Database of Institut Paoli-Calmettes patients diagnosed with cardia cancer

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cardia cancer

Exclusion Criteria:

-

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Cardia Cancer
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2002-01; Primary Completion 2030-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Survival of patients | 10 years
  Overall survival of all patients who come in the center

SECONDARY OUTCOMES:
Collection of patients characteristics | 10 years
  Collection of characteristics of patients treated at Institut Paoli Calmettes in order to set up prospective and retrospective studies

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli-Calmettes, Marseille, Bouches-du Rhône, France

IPD SHARING:
Plan to Share IPD: No